CLINICAL TRIAL: NCT00073398
Title: A Phase I/II Study of Tergenpumatucel-L (HyperAcute Lung) an Antitumor Vaccination Using Alpha (1,3) Galactosyltransferase Expressing Allogeneic Tumor Cells in Patients With Refractory or Recurrent Non-Small Cell Lung Cancer
Brief Title: Vaccine Treatment for Advanced Non-Small Cell Lung Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: NewLink Genetics Corporation (Industry)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: Lumos Pharma (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NLG0101; 04-C-0049; NCT00075790 (obsolete NCT alias)
Record Dates: First submitted 2003-11-19; First posted 2003-11-20 (Estimated); Last update posted 2020-05-28 (Actual); Status verified 2020-05

CONDITIONS: Non-small Cell Carcinoma; Adenocarcinoma of Lung; Squamous Cell Carcinoma; Large Cell Carcinoma; Lung Neoplasms
Keywords: Anti-tumor Vaccination; Alpha (1,3) Galactosyltransferase; Allogeneic Tumor Cells; Hyperacute Lung; NSCLC; Lung Cancer; Non-Small Cell Lung Cancer
MeSH Terms: conditions — Adenocarcinoma of Lung; Carcinoma, Squamous Cell; Carcinoma, Large Cell; Lung Neoplasms; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental): Ph II Arm 1
  Interventions: Biological: Drug: Hyperacute Lung Cancer Cell Vaccine

INTERVENTIONS:
Biological: Drug: Hyperacute Lung Cancer Cell Vaccine — At dose levels I IV the vaccine cells will be injected intradermally every four weeks for four cycles. Dosage will vary from a total of 3 x 106 to 100 x 106 HyperAcute -Lung Cancer Vaccine cells administered per vaccination cycle. At dose level V patients will receive injections of the HyperAcute -Lung Cancer Vaccine cells to include one (1) initial priming vaccine dose of 500 x 106 cells followed by seven (7) booster vaccine cell doses of 300 x 106 HyperAcute -Lung Cancer cell vaccine cells every two weeks. In Phase II, patients will receive 300 x 106 HyperAcute -Lung Cancer cell vaccine cells every two weeks for a total of 8 doses (4 months).

SUMMARY:
This 2-phase study will determine the safety of treating patients with non-small cell lung cancer with the genetically engineered HyperAcute-Lung cancer vaccine. It will establish the proper vaccine dose and will examine side effects and potential benefits of the treatment. The vaccine contains killed lung cancer cells containing a mouse gene that causes the production of a foreign pattern of protein-sugars on the cell surface. It is hoped that the immune response to the foreign substance will stimulate the immune system to attack the patient's own cancer cells that have similar proteins without this sugar pattern, causing the tumor to remain stable or shrink.

Patients 18 years of age or older with non-small cell lung cancer that has recurred or no longer responds to standard treatment may be eligible for this study. Candidates will be screened with a medical history and physical examination, blood tests, urinalysis, chest x-rays, and lung function testing. CT, MRI, PET, and ultrasound scans of the chest may be obtained if needed.

Participants will receive four vaccinations a month apart from each other. The vaccines will be injected under the skin, similar to the way a tuberculosis skin test is given. Phase I of the study will treat successive groups of patients with increasing numbers of the vaccine cells to evaluate side effects of the treatment and determine the optimum dose. Phase II will look for any beneficial effects of the vaccine given at the highest dose found to be safe in Phase I. Weekly blood samples will be drawn during the 4 months of vaccine treatment. In addition, patient follow-up visits will be scheduled every 2 months for the first year after vaccination and then every 3 months for the next 2 years for the following tests and procedures to evaluate treatment response and side effects:

* Medical history and physical examination
* Blood tests
* X-rays and various scans (nuclear medicine/CT/MRI)
* FACT-L Assessment questionnaire to measure the impact of treatment on the patient's general well-being. The questionnaire is administered before beginning treatment, before each vaccination, and during follow-up visits after completing the treatment. It includes questions on the severity of lung cancer symptoms and the ability to perform normal activities of daily life.

In addition to the above procedures, 3 skin punch biopsies will be done at the vaccination site to look for a local immune response. For this procedure, an area of skin is numbed with an anesthetic and a 4 mm (about 1/4-inch) circular area is removed, using a sharp cookie cutter-type instrument. Also, one blood sample per year will be collected for the next 15 years to monitor the safety of the gene transfer. Patients whose lung cancer spreads to the skin, superficial soft tissues, or a superficial lymph node may be asked to undergo a biopsy of the lesion to see what effect the treatment may be having on the tumor.

DETAILED DESCRIPTION:
Background:

* Lung cancer remains the leading cause of cancer death with an estimated 174,400 new cases and 162,400 deaths each year in the U.S.
* Despite attempts at early diagnosis and the development of new therapeutic agents, there has been only limited improvement in the outcome for patients with advanced lung cancer.
* A enzyme called alpha(1,3)galactosyltranferase (alphaGT) that is not found in humans can transfer sugars on to proteins in human cells that can make them highly immunogenic and cause them to be rejected by the body.
* Antitumor vaccination using killed donor human lung cancer cells expressing alphaGT may stimulate immune responses in patients against their own lung cancer because their lung cancer may share antigens with the vaccine cells that have been made more immunogenic by expression of alphaGT.

Objectives:

Phase I has been completed.

Phase II

* To assess the tumor response rate of anti-tumor vaccination using irradiated allogeneic lung cancer cell lines genetically engineered to express the murine alpha(1,3)galactosyltransferase enzyme in patients with advanced, recurrent or refractory non-small cell lung cancer.
* To assess the immunological response of patients with lung cancer undergoing antitumor vaccination with irradiated allogeneic lung cancer cell lines genetically engineered to express murine alpha(1,3)galactosyltransferase.
* Assess the survival distribution as well as the duration of response.

Eligibility:

* Non-small cell lung cancer (Adenocarcinoma, squamous cell carcinoma, large cell anaplastic carcinoma and bronchoalveolar carcinoma).
* Stage IV, recurrent or treatment refractory disease.
* No exclusion for prior therapy. Prior therapy may include surgery, radiation, immunotherapy, and chemotherapy regimens. EGFR inhibitors or monoclonal antibodies are included as chemotherapy.
* Patients must have a granulocyte count of greater than or equal to 1000/microL, platelets greater than or equal to 100,000/microL, hemoglobin greater than 10.0 gm/dL, albumin greater than or equal to 3.0 gm/dL and acceptable hepatic and renal function.
* No systemic corticosteroids.

Design (Phase II):

* Patients will be intradermally vaccinated with 300 million alpha(1,3)galactosyltranferase-expressing vaccine cells every 2-weeks to complete a total of eight vaccinations.
* Patients will be monitored for tumor and immunological responses and safety.

ELIGIBILITY:
* Phase II Eligibility Criteria

Must be confirmed within 4-weeks of vaccination except for Beta-HCG (confirm within 1-week) when appropriate. Tumor measurements must be performed within 2-weeks of enrollment.

INCLUSION CRITERIA:

Histological diagnosis of non-small cell lung cancer (NSCLC). Squamous cell (epidermoid), adenocarcinoma, bronchoalveolar carcinoma and large cell anaplastic lung carcinoma histologies are eligible. Mixed histologies of NSCLC (i.e., adenosquamous) are eligible. Mixed NSCLC/small cell lung carcinoma (SCLC), and variant large and small cell lung cancer are NOT eligible for this study.

Patients being treated at the NCI must have their pathology reviewed and confirmed by the NCI Laboratory of Pathology. Patients being treated at MCG must have their pathology reviewed and confirmed by the MCG Pathology Department.

Metastatic (AJCC Stage IV- any T, any N, M1), progressive, recurrent or refractory NSCLC. Patients may not be eligible for other curative intent treatment (e.g., surgical resection).

For the purpose of eligibility for this trial, the above-cited disease states are defined as follows:

Progressive NSCLC- Defined as increasing measurable disease or the appearance of new measurable disease by RECIST criteria despite treatment.

Recurrent NSCLC- Defined as the re-appearance of measurable disease or the appearance of new measurable disease by RECIST criteria after prior successful treatment or complete response.

Refractory NSCLC- Defined as achieving less than a complete response and having residual measurable by RECIST criteria after prior treatment with chemotherapy, targeted or small molecules, monoclonal antibodies or any combination of these.

Eastern Cooperative Oncology Group (ECOG) Performance Status less than or equal to 2.

Serum albumin greater than or equal to 3.0 gm/dL.

Expected survival greater than or equal to 4 months.

Adequate organ function including:

* Marrow: Hemoglobin greater than or equal to 10.0 gm/dL, absolute granulocyte count (AGC) greater than or equal to 1,000/mm(3) platelets greater than or equal to 100,000/mm(3), absolute lymphocyte count greater than or equal to 475/mm(3).
* Hepatic: Serum total bilirubin less than or equal to 1.5 times the upper limit of normal (ULN) with the exception of less than 2.9 mg/dL for patients with Gilbert's disease, ALT (SGPT) and AST (SGOT) less than or equal to 2.5 times the ULN.
* Renal: Serum creatinine (sCr) less than or equal to 1.5 times the upper limit of normal, or creatinine clearance (Ccr) greater than or equal to 50 mL/min.

All On-Study Tests must be less than or equal to CTC Grade I toxicity for patients to be eligible for study, excluding serum LDH levels. PT, PTT must be less than or equal to 1.5 times ULN except for patients who are on therapeutic anticoagulant therapy.

Measurable disease as defined by RECIST Criteria.

Subjects must have negative serologies for hepatitis viruses B and C, and HIV prior to entering study.

Prior therapy for NSCLC that may include surgery, radiation therapy, immunotherapy, and/or prior chemotherapy regimens (including neoadjuvant and adjuvant treatment). There are no restrictions to the number of prior therapies subjects have received.

Treatment with a single course of gefitinib or (Iressa), or erlotinib (Tarceva), or other small molecule or targeted therapies, or monoclonal antibody therapy will be considered and count as prior chemotherapy.

Patients that refuse chemotherapy are eligible.

Patients must be greater than or equal to 4 weeks since major surgery, radiotherapy, chemotherapy (6-weeks if they were treated with a nitrosourea or mitomycin) or biotherapy/targeted therapies and recovered from the toxicity of prior treatment to less than or equal to CTC grade 1, exclusive of alopecia or fatigue.

Patients must have the ability to understand the study, its risks, side effects, potential benefits and be able to give written informed consent to participate. Patients may NOT be consented by a durable power of attorney (DPA).

Male and female subjects of child producing potential must agree to use contraception or avoidance of pregnancy measures while enrolled on study and receiving the experimental drug, and for one month after the last immunization.

Patients should have sites of NSCLC that are accessible to needle, punch or other limited biopsy, be at low risk for biopsy and be willing to undergo tumor core needle biopsy, punch or other similar biopsy pre-vaccination and again post-vaccination. Such sites may include skin and soft tissue metastases, adrenal gland metastases, peripheral lymph nodes (supraclavicular, axillary, or inquinal), a pulmonary lesion at low risk for complications defined as lesions greater than 1.5 cm surrounded by aerated lung, pleural based masses greater than 1.5 cm and lesions not associated with a major pulmonary vessel, or other disease sites that may undergo biopsy with minimal discomfort and risk to the patient. These biopsies are optional.

EXCLUSION CRITERIA:

Age less than 18-years-old.

Active CNS metastases or carcinomatous meningitis.

Hypercalcemia greater than 2.9 mmol/L, unresponsive to standard therapy (e.g., I.V. hydration, diuretics, calctonin and/or bisphosphate therapy).

Pregnant or nursing women due to the unknown effects of vaccination on the developing fetus or newborn infant.

Other malignancy within five years, unless the probability of recurrence of the prior malignancy is less than 5%. Patient's curatively treated for squamous cell carcinoma and basal cell carcinoma of the skin and carcinoma in situ of the uterine cervix (CIN) or patients with a history of malignant tumor in the past that have been disease free for at least five years are also eligible for this study.

History of organ transplant, or current active immunosuppressive therapy (such as cyclosporine, tacrolimus, etc.).

Subjects taking systemic corticosteroid therapy for any reason including replacement therapy for hypoadrenalism, are not eligible. Subjects receiving inhaled or topical corticosteroids are eligible. Subjects who require systemic corticosteroids after beginning vaccinations, will be removed from the study.

Significant or uncontrolled congestive heart failure (CHF), myocardial infarction, significant ventricular arrhythmias within the last six months or significant pulmonary dysfunction.

Active infection or antibiotics within 1-week prior to study, including unexplained fever (Temp. greater than 38.1 degrees C).

Autoimmune disease (e.g., systemic lupus erythematosis, active rheumatoid arthritis, etc) with the exception of vitiligo. Patients with a remote history of asthma or mild active asthma are eligible.

Other serious medical conditions that may be expected to limit life expectancy to less than 2-years (e.g., liver cirrhosis).

Any condition, psychiatric or otherwise, that would preclude informed consent, consistent follow-up or compliance with any aspect of the study (e.g., untreated schizophrenia or other significant cognitive impairment, etc).

A known allergy to any component of the alpha(1,3)galactosyltransferase tumor vaccine or cell lines from which it is derived.

Patients having undergone splenectomy or prior vaccine therapy for their NSCLC.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2003-11; Primary Completion 2012-11 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Safety and response rate | Days 57, 85, 127

CONTACTS AND LOCATIONS:
Overall Officials: Arun Rajan, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Pruitt SK, Kirk AD, Bollinger RR, Marsh HC Jr, Collins BH, Levin JL, Mault JR, Heinle JS, Ibrahim S, Rudolph AR, et al. The effect of soluble complement receptor type 1 on hyperacute rejection of porcine xenografts. Transplantation. 1994 Feb;57(3):363-70. doi: 10.1097/00007890-199402150-00009. PMID 8108871
- [Background] Lai L, Kolber-Simonds D, Park KW, Cheong HT, Greenstein JL, Im GS, Samuel M, Bonk A, Rieke A, Day BN, Murphy CN, Carter DB, Hawley RJ, Prather RS. Production of alpha-1,3-galactosyltransferase knockout pigs by nuclear transfer cloning. Science. 2002 Feb 8;295(5557):1089-92. doi: 10.1126/science.1068228. Epub 2002 Jan 3. PMID 11778012
- [Background] Galili U, Shohet SB, Kobrin E, Stults CL, Macher BA. Man, apes, and Old World monkeys differ from other mammals in the expression of alpha-galactosyl epitopes on nucleated cells. J Biol Chem. 1988 Nov 25;263(33):17755-62. PMID 2460463
- See also: NIH Clinical Center Detailed Web Page — http://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2004-C-0049.html